CLINICAL TRIAL: NCT01026857
Title: Phase II, Parallel-group, Placebo Controlled, Double-blind, Randomised, Multicenter Study to Investigate the Efficacy of Two Dosages of Propionyl-L-Carnitine Colon Release Tablets in Patients Affected by Ulcerative Colitis Under Oral Stable Treatment
Brief Title: Propionyl-L-Carnitine in Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: sigma-tau i.f.r. S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ST261 DM 01 004
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2009-12

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PLC Colon release tablet 1 g (Experimental): 40 patients each arm
  Interventions: Drug: Propionyl-L-Carnitine; Drug: Placebo
- PLC colon release tablet 2 g (Experimental): 40 patients each arm
  Interventions: Drug: Propionyl-L-Carnitine; Drug: Placebo
- Placebo PLC colon release tablet 2 g (Placebo Comparator): 40 patients each arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propionyl-L-Carnitine — PLC colon release tablet 1 g/die for 4 weeks
  Other Names: Dromos
  Arms: PLC Colon release tablet 1 g
Drug: Propionyl-L-Carnitine — PLC colon release tablet 2 g/die for 4 weeks
  Other Names: Dromos
  Arms: PLC colon release tablet 2 g
Drug: Placebo — Placebo PLC colon release tablet 2 g/die for 4 weeks

SUMMARY:
The purpose of this study is to determine whether Propionyl-L-carnitine administration may ameliorate the illness in patients affected by mild to moderate ulcerative colitis already in treatment with one of the standard treatments (corticosteroids excluded).

DETAILED DESCRIPTION:
The trial foresees the administration of 2 different dosages of Propionyl-L-carnitine (ST261) colon release tablets, 1 g/die and 2 g/die. The primary objective of this trial is to evaluate the clinical/endoscopic response defined as a lowering of the Disease Activity Index (DAI score) of at least 3 points ot the reaching of remission, the clinical/endoscopic remission (DAI score <= 2 with no individual subscore > 1) and histological efficacy of the two combined dosages of PLC (i.e. PLC 1 g/die + 2 g/die) in comparison to placebo, defined as an improvement of the Histological Index (HI) of at least 1 point at the end of the study (a final HI score of <= 1 will be defined as an histological remission).

The secondary objective is to evaluate the clinical/endoscopic and histological efficacy of the two dosages of PLC individually considered in comparison to Placebo, in order to gather information on the dosage to be used in subsequent trials. The safety and tolerability of the regimens studied will also be objectives of the study.

ELIGIBILITY:
Inclusion Criteria:

* Have read the Information for the Patient and signed the Informed Consent Form.
* Age comprised between 18 and 75 included.
* If female, not pregnant or nursing.
* For women of childbearing potential, willingness to avoid a pregnancy during the treatment period and for at least 1 month from the last dose of drug.
* Availability of a pancolonoscopy and histology both confirming the diagnosis of active ulcerative colitis.
* Disease Activity Index comprised between 3 and 10, inclusive, (mild to moderate ulcerative colitis).
* On one of the following treatments for ulcerative colitis prior to baseline visit:

  1. Stable background oral aminosalicylates (mesalazine, balsalazide, olsalazine) or sulfasalazine therapy for greater than or equal to 4 weeks prior to baseline assessments.
  2. Stable background mercaptopurine or azathioprine for greater than or equal to 12 weeks prior to baseline assessments.

Exclusion Criteria:

* First diagnosis of ulcerative colitis.
* Crohn's disease.
* Current or previous (in the last 10 days preceding the screening) use of systemic corticosteroids.
* Use of antibiotics in the last 10 days preceding the screening.
* Use of NSAID's in the last 10 days preceding the screening.
* Use of probiotics in the last 10 days preceding the screening
* Positive stool culture (when performed, according to Investigator's judgment, to assess possible parasitologic infection(s)).
* Significantly impaired liver, renal, pulmonary or cardiovascular function.
* History of colon resection.
* Diverticulitis.
* Diagnosis of proctitis
* Stable rectally administered therapy in the last 10 days.
* Active or chronic infection(s).
* Simultaneous participation in another clinical trial, or participation in any clinical trial involving investigational drugs within 3 months from enrolment into the present study.
* Any physical or psychological condition in a patient that could let the investigator suspect his/her poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2006-05; Primary Completion 2009-04 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Disease Activity Index score | baseline, week 4

SECONDARY OUTCOMES:
Adverse Events | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni B. Gasbarrini, M.D., Principal Investigator — Policlinico Universitario "A. Gemelli" - Rome - Italy; Gabriele Bianchi Porro, M.D., Principal Investigator — Ospedale "L. Sacco" - Milan - Italy; Agesilao D'Arienzo, M.D., Principal Investigator — A.O. Universitaria Federico II - Naples - Italy; Daniela Valpiani, M.D., Principal Investigator — P.O. Morgagni Pierantoni - Forlì - Italy; Maurizio Koch, M.D., Principal Investigator — Ospedale "S. Filippo Neri" - Rome - Italy; Ewa Malecka-Panas, M.D., Principal Investigator — Klinika Przewodu Pokarmowego Szpital Kliniczny Nr 1 - Lodz - Poland; Leszek Paradowski, M.D., Principal Investigator — Samodzielny Publiczny Szpital Kliniczny Nr 3 - Wroclaw - Poland; Konrad Lesniakowski, M.D., Principal Investigator — Wojewodzki Szpital - Wroclaw - Poland; Limas Kupcinskas, M.D., Principal Investigator — Kaunas Medical University Clinic - Kaunas - Lithuania; Goda Denapiene, M.D., Principal Investigator — Vilnius University Santariskiu Hospital - Vilnius - Lithuania; Vladimir B. Grinevich, M.D., Principal Investigator — State Institution "Regional Military Clinical Hospital N°422 named after Solovyov of Ministry of Defence of Russia - Saint Petersburg - Russia; Elena Sishkova, M.D., Principal Investigator — Federal State Healthcare Institution "Clinical Hospital N°122 named after L.G. Sokolov of Federal Medical and Biological Agency" - Saint Petersburg - Russia; Konstantin P. Zhidkov, M.D., Principal Investigator — St Petersburg State Healthcare Institution "Municipal Hospital N°26" - Saint Petersburg - Russia; Igor G. Bakulin, M.D., Principal Investigator — Federal State Institution "7th Central Military Clinical Aviation Hospital of Ministry of Defence of Russia" - Moscow - Russia; Tatiana L. Mikhailova, M.D., Principal Investigator — Federal State Institution "State Scientific Centre of Coloproctology of Rosmedtechnologij" - Moscow - Russia
Locations (15):
- Italy (5):
  - Hospital Morgagni - Pierantoni, Forlì
  - Ospedale "L. Sacco", Milan
  - University Federico II, Naples
  - Hospital S. Filippo Neri, Rome
  - Policlinico "A. Gemelli", Rome
- Lithuania (2):
  - Kaunas Medical University Clinic, Kaunas
  - Vilnius University Santariskiu Hospital, Vilnius
- Poland (3):
  - Klinika Przewodu Pokarmowego Szpital Kliniczny Nr 1, Lodz
  - Samodzielny Publiczny Szpital Kliniczny Nr 3 Katedra i Klinika Gastroenterologii AM, Wroclaw
  - Wojewódzki Szpital Specjalistyczny Klinika Gastroenterologii, Wroclaw
- Russia (5):
  - Federal State Institution "7-th Central Military Clinical Aviation Hospital of Ministry of Defence of Russia", Moscow
  - Federal State Institution "State Scientific Centre of Coloproctology of Rosmedtechnologij", Moscow
  - State Institution "Regional Military Clinical Hospital № 442 named after Z.P. Solovyov of Ministry of Defence of Russia", Saint Petersburg
  - Federal State Healthcare Institution "Clinical Hospital № 122 named after L.G. Sokolov of Federal Medical and Biological Agency", Saint Petersburg
  - St-Petersburg State Healthcare Institution "Municipal Hospital № 26", Saint Petersburg

REFERENCES:
- [Derived] Mikhailova TL, Sishkova E, Poniewierka E, Zhidkov KP, Bakulin IG, Kupcinskas L, Lesniakowski K, Grinevich VB, Malecka-Panas E, Ardizzone S, D'Arienzo A, Valpiani D, Koch M, Denapiene G, Vago G, Fociani P, Zerbi P, Ceracchi M, Camerini R, Gasbarrini G. Randomised clinical trial: the efficacy and safety of propionyl-L-carnitine therapy in patients with ulcerative colitis receiving stable oral treatment. Aliment Pharmacol Ther. 2011 Nov;34(9):1088-97. doi: 10.1111/j.1365-2036.2011.04844.x. Epub 2011 Sep 19. PMID 21929562